CLINICAL TRIAL: NCT03328234
Title: A Randomized Phase III Study of Simultaneous Integrated Boost Intensity Modulated Radiation Therapy (SIB-IMRT) With or Without Concurrent Chemotherapy Followed by Consolidation Chemotherapy for Extensive Lymphatic Metastasis of Esophageal Cancer - 3JECROG-P03
Brief Title: Radiotherapy With or Without Concurrent Chemotherapy for Extensive Lymphatic Metastasis of Esophageal Cancer - 3JECROG P-03
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Zefen Xiao, Pricipal investigator, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 3JECROG P-03
Record Dates: First submitted 2017-10-28; First posted 2017-11-01 (Actual); Last update posted 2019-01-02 (Actual); Status verified 2018-12

CONDITIONS: IMRT With or Without Concurrent Chemotherapy for Esophageal Cancer
MeSH Terms: interventions — Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SIB-IMRT combined chemotherapy with IFI (Experimental)
  Interventions: Radiation: SIB-IMRT; Drug: Paclitaxel; Drug: Platinum-Based Drug; Other: Involved Field Irradiation (IFI)
- SIB-IMRT with IFI (Experimental)
  Interventions: Radiation: SIB-IMRT; Drug: Paclitaxel; Drug: Platinum-Based Drug; Other: Involved Field Irradiation (IFI)

INTERVENTIONS:
Radiation: SIB-IMRT — Patients receive radiotherapy once daily, 5 days a week for an average of 5.5 weeks. Radiotherapy is delivered to achieve a prophylactic dosage of 50.4Gy to PTV and 59.92Gy to PGTV in 28 fractions, respectively.
Drug: Paclitaxel — 45-50mg/m2, once a week, concurrent with radiotherapy for 5-6weeks
  Arms: SIB-IMRT combined chemotherapy with IFI
Drug: Platinum-Based Drug — Nedaplatin or Lobaplatin or Cisplatin, 20-25mg/m2, once a week, concurrent with radiotherapy for 5-6weeks
  Arms: SIB-IMRT combined chemotherapy with IFI
Drug: Paclitaxel — 135-150mg/m2 on day1,every 3 weeks, 2 cycles, 1 month after completion of radiotherapy
Drug: Platinum-Based Drug — Nedaplatin or Lobaplatin or Cisplatin, 50-80mg/m2 on day1 (Lobaplatin,50mg on day1 ),every 3 weeks, 2 cycles, 1 month after completion of radiotherapy
Other: Involved Field Irradiation (IFI) — CTV was defined as GTV with a 3.0-5.0 cm craniocaudal margin and a 0.6-0.8 cm lateral margin and GTVnd with a 0.5-1.0 cm margin.

SUMMARY:
The investigators aimed to compare elective nodal irradiation versus involved field irradiation with or without concurrent chemotherapy and the addition of consolidation chemotherapy for patients with extensive lymphatic metastasis of esophageal cancer.

ELIGIBILITY:
Inclusion Criteria:

* Age<70
* Diagnosis of clinical stage T2-4N0-1M1（According to UICC 2002）
* A untreated squamous esophageal carcinoma
* Karnofsky performance status(KPS)≥ 70 and Charlson score ≤3
* Adequate organ function
* No known history of drug allergy
* Blood routine examination : WBC≥4.0
* hepatic and renal function are normal

Exclusion Criteria:

* Age≥ 70 or ≤ 16
* Already received the treatment of chemotherapy or radiotherapy
* Pregnant or lactating females
* Known drug allergy
* Without agreement of informed consent form
* Insufficient hepatorenal function or Blood routine examination
* Severe cardiovascular diseases, diabetes with uncontrolled blood sugar, mental disorders, uncontrolled severe infection, active ulceration which need intervention.

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Estimated)
Dates: Start 2017-09-01 (Actual); Primary Completion 2021-08-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall survival (OS) | 1 year
Overall survival (OS) | 2 year
Overall survival (OS) | 3 year

SECONDARY OUTCOMES:
Progression-free survival (PFS) | 1 year
Progression-free survival (PFS) | 2 year
Progression-free survival (PFS) | 3 year
Local recurrence-free rate（LRFS） | 1 year
Local recurrence-free rate（LRFS） | 2 year
Local recurrence-free rate（LRFS） | 3 year
Completion Rate | up to 2 year
Adverse events | up to 5 year

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Radiation Oncology, Cancer Hospital, National Cancer Center, Chinese Academy of Medical Sciences (CAMS) and Peking Union Medical College (PUMC), Beijing, China